CLINICAL TRIAL: NCT06039475
Title: Risk Factors Associated With High Altitude Sickness: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sishir Poudel, Doctor, B.P. Koirala Institute of Health Sciences
Other Study IDs: 339/2023
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Acute Mountain Sickness; High Altitude Pulmonary Edema; High Altitude Cerebral Edema
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with AMS/HACE/HAPE
- Control: Healthy Individuals

SUMMARY:
Research Title: RISK FACTORS ASSOCIATED WITH HIGH ALTITUDE SICKNESS: A CASE-CONTROL STUDY Rationale: The Study will help us to identify risk factors of high altitude sickness among Nepalese and International patients.

Aims and Objectives:

* To identify risk factors for high altitude sickness, including AMS, HACE, and HAPE.
* To compare the prevalence of high altitude sickness between individuals who ascended rapidly versus those who ascended slowly.
* To examine the association between high altitude sickness and various demographic and environmental factors, such as age, sex, altitude, and temperature.
* To evaluate the effectiveness of preventative measures, such as gradual ascent and medication, in reducing the risk of high altitude sickness Research Hypothesis (if relevant): N/A

  1. Material & Methods:

     1. Whether study involves Human/animals or both : Human
     2. Population/ participants: Patients presenting in Emergency Ward of District Hospital, Mustang with AMS (Acute Mountain Sickness), HAPE (High altitude Pulmonary Oedema) or HACE (High altitude Cerebral Oedema) as CASES Healthy volunteers who didn't develop any symptoms of AMS/HAPE/HACE after their trip to high altitude as CONTROLS
     3. Type of study design: : Case Control Study
     4. Human study :

        Inclusion Criteria: Cases: Individuals age 18 years or older who have been diagnosed with AMS based on a LLS score of ≥3 or HAPE or HACE.

        Controls: Individuals age 18 years or older who did not develop AMS during their trip to high altitude as the cases, and who are matched to cases on age and sex.

        Exclusion Criteria:
        * Those who deny consent for participation.
        * Age<18 years
        * Pregnant Women
     5. Expected sample size :

        Sample size calculation: Mentioned in methodology
     6. Control groups : N/A
     7. Probable duration of study: 180 days
     8. Setting: Emergency Ward
     9. Parameter/Variables to be applied/measured Independent Variables i. Socio-demographic characteristics such as age, sex, address, nationality.

     Dependent Variables:

     i. Symptoms of Presentation ii. Ascent Rate iii. Co-morbidities iv. Past History including previous history of altitude sickness v. Personal History such as smoking, alcohol intake, recreational drugs vi. Awareness on High Altitude Sickness vii. Intake of Prophylactic medicine (Acetazolamide) viii. Past history of Covid-19 , TB

     Outcome measures:

     Primary (main outcome): All dependent variables

     (i) Rational for statistical methods to be employed : Data will be entered in Microsoft Excel and converted it into SPSS for statistical analysis .

     Descriptive statistics will be used to summarize the characteristics of cases and controls. Univariate and multivariate logistic regression analyses will be performed to assess the association between risk factors and high altitude sickness. The results will be reported as odds ratios with corresponding 95% confidence intervals. A p-value of less than 0.05 will be considered statistically significant.

     (ii) Ethical clearance : Ethical clearance will be obtained from National Health Research Council of Nepal (iii) Permission to use copyright questionnaire/Pro forma: Not applicable

     (j) Maintain the confidentiality of subject Confidentiality of the participants will be maintained. Whether available resources are adequate: Yes
     1. Other resources needed: No
     2. For Intervention trial: Not applicable

DETAILED DESCRIPTION:
INTRODUCTION

The primary environmental factor at high elevations is a decrease in barometric pressure. This decrease leads to a reduction in the partial pressure of oxygen at each stage of the process that carries oxygen from the air to the cells' mitochondria. This hypobaric hypoxia initiates a sequence of physiological responses that generally enable an individual to endure and adjust to the low-oxygen environment. However, there are instances where these responses become maladaptive, resulting in one of three forms of acute altitude illness: acute mountain sickness (AMS), high-altitude cerebral oedema (HACE), and high-altitude pulmonary oedema (HAPE). These diseases may occur within several hours or up to 5 days after ascending to a particular height and can range in severity from mild, having minimal impact on the scheduled travel itinerary, to a life-threatening condition..(1) Acute mountain sickness (AMS) is characterized by non-specific symptoms that emerge at altitudes of ⩾2500 m among unacclimatized individuals. These symptoms usually appear with a delay of 4-12 hours after arriving at a new altitude, and tend to be most intense after the first night spent there. When appropriate measures are taken, these symptoms typically resolve on their own.(2) Acute mountain sickness (AMS) is a collection of symptoms that typically involves a headache and at least one other symptom such as nausea/vomiting, fatigue, dizziness, or difficulty sleeping. It usually appears 6-12 hours after arriving at high altitude and generally resolves within 1-3 days. If left untreated, AMS can progress to high-altitude cerebral edema (HACE), which is characterized by altered mental status such as impaired mental capacity, drowsiness, stupor, and ataxia. Coma and even death can occur as soon as 24 hours after these symptoms develop.(3) High altitude pulmonary edema (HAPE) is a type of pulmonary edema that is non-cardiogenic in nature and may not be preceded by acute mountain sickness. Typically, it occurs between one and four days after arriving at altitudes higher than 2500 m.(4) There are several risk factors associated with altitude sickness, including the elevation of the individual's home, maximum altitude, sleeping altitude, rate of ascent, latitude, age, gender, physical condition, intensity of exercise, pre-acclimatization, genetic make-up, and pre-existing diseases. Both men and women are at similar risk of developing AMS, although some studies suggest that women may be slightly more susceptible. Contrary to popular belief, older individuals do not appear to be at higher risk of AMS. In fact, some studies suggest that younger individuals may be more susceptible. A previous history of AMS is a significant predictor for developing AMS upon subsequent exposure to comparable altitudes(5) It is unclear if other factors such as age, obesity, gender, level of fitness, and nicotine or alcohol consumption are significant risk factors for altitude sickness in mountaineering populations. The primary determinants of AMS appear to be the level of acclimatization, rate of ascent, and individual susceptibility. Further research is needed to fully understand the impact of these additional factors on the development of altitude sickness in mountaineering populations.(6) Meta-analyses of observational field studies have demonstrated that prophylactic acetazolamide can reduce the symptoms of acute mountain sickness. The drug is typically prescribed at doses between 125 mg and 1 g per day, with most patients receiving 125 mg or 250 mg twice daily. However, it is important to note that acetazolamide does not prevent the symptoms of acute mountain sickness when an individual ascends too quickly.(7) The Mustang study site is known for its several high-altitude attractions, including the world-renowned Thorong La Pass (5416m) in the Annapurna trekking circuit, the Muktinath Temple (3800m), Lo Manthang (3840m), and the Kora La Pass (4660m). In recent years, improvements to major roadways have increased connectivity to these attractions, resulting in an increased flow of visitors and shorter travel times. However, this has also led to a higher likelihood of individuals rapidly ascending from lower elevations to a hypobaric hypoxia environment, thereby increasing the risk for developing high-altitude illness during the initial few days of travel.(8)

LITERATURE REVIEW In a study done among trekkers climbing a 5400 m high pass in the Nepalese Himalaya the overall prevalence of AMS was 63%. AMS was positively correlated with rate of ascent and negatively correlated with pre-trek acclimatization. Women suffered more frequently and more seriously from AMS. Body mass index (weight/length2) was significantly correlated with AMS in men. No significant association was found between AMS and age, smoking habits, use of oral contraceptives, previous high altitude experience, special pre-trek training, size of trekking party or whether the trek was agency- or self-organised. Of trekkers, 80% had elementary knowledge of the diagnosis and treatment of AMS.(9) In a one-year study conducted at Mustang District Hospital, it was found that approximately one-fourth (25.7%) of the 105 patients exhibiting symptoms were not meeting the criteria of LLS to be classified as AMS patients. Out of the remaining three-fourths (74.3%) who were diagnosed with AMS, 61.5% had mild symptoms, 35.9% had moderate symptoms, and only 2.6% had severe symptoms. In the dataset, there was only one case of HACE and two cases of HAPE. Among patients with AMS, approximately 73.1% reported experiencing gastrointestinal symptoms, 84.6% reported dizziness, and a majority of 97.4% reported fatigue. Ascent rate was strongly associated with the likelihood of developing severe AMS among travellers with AMS symptoms.(10) A preliminary study sponsored by the Himalayan Rescue Association of AMS among pilgrims to a holy lake (Gosaikunda) at 4154 m in Nepal, revealed that out of 5163 pilgrims who came to the lake, 229 (4.4%) developed AMS. The severity of the illness correlated with the rapidity of ascent, but there was no difference in severity between men and women.(11) A study was conducted in a total of 162 mountaineers (assuming that the more experienced mountaineers of the Western Alps are less susceptible to developing AMS than recreational mountaineers of the Eastern Alps or tourist populations), 79 in the Eastern Alps (3454 m) and 83 in the Western Alps (3817 m) on the morning after their first night at high altitude. A diagnosis of AMS was based on a Lake Louise Scoring, thirty of 79 subjects (38.0%) suffered from AMS at 3454m in the Eastern Alps as did 29 of 83 (34.9%) at 3817m in the Western Alps. After adjustment for altitude, the prevalence in the Western Alps constituted 24.5%, which differed significantly (p=0.04) from that found in the Eastern Alps. The lower mountaineering experience of mountaineers in the Eastern Alps turned out to be the only factor for explaining their higher AMS prevalence.(12) A study was done on 27 mountaineers on the day of arrival at the Capanna Margherita (4559 m) and on the next morning. Susceptibility was assessed based on previous AMS episode and pre exposure was defined as having spent more than 4 d above 3000 m during the 2 months preceding the climb to the Capanna Margherita. Slow ascent was defined as ascending in more than 3 d. In susceptible individuals, the prevalence of AMS was 58% with rapid ascent and no preexposure, 29% with preexposure only, 33% with slow ascent only, and 7% with both preexposure and slow ascent. The corresponding values for nonsusceptible individuals were 31%, 16%, 11%, and 4%. The overall odds ratio for developing AMS in susceptible versus nonsusceptible individuals was 2.9 (95% confidence interval, 2.1- 4.1). Age, gender, training, body mass index, alcohol intake, and cigarette smoking had no significant effect in bivariate analyses or in multivariate logistic regressions. In conclusion individual susceptibility, rate of ascent, and preexposure are the major, independent determinants for prevalence of AMS.(6) In a meta-analysis done studying acetazolamide for the prevention of AMS, when all of the reported symptoms were pooled together, the average ES was -0.38, indicating that drug prophylaxis was effective in reducing the most common symptoms of AMS. When examined individually, the ES for preventing headache was -0.54, nausea was -0.29, and insomnia was -0.42.(7)

RESEARCH AIM AND OBJECTIVES Primary Objective: To identify risk factors for high altitude sickness, including AMS, HACE, and HAPE

Specific Primary Objectives:

To compare the prevalence of high altitude sickness between individuals who ascended rapidly versus those who ascended slowly.

To examine the association between high altitude sickness and various demographic and environmental factors, such as age, sex, altitude, and temperature.

To evaluate the effectiveness of preventative measures, such as gradual ascent and medication, in reducing the risk of high altitude sickness

METHODOLOGY

4. Research Design and Methodology 4.1 Research Method: Case Control Study

Study Variables:

Socio-demographic characteristics such as age, sex, address including altitude and nationality.

Symptoms of Presentation, Ascent Rate, Co-morbidities, Past History including COVID,TB previous history of altitude sickness, Personal History such as smoking, alcohol intake, Awareness on High Altitude Sickness and Intake of Prophylactic medicine (Acetazolamide)

Outcome variables: All dependent variables 4.3 Study Design (Specify): Case Control Study 4.4 Study Site and Its Justification: MUSTANG DISTRICT HOSPITAL 4.5 Study Population (Specify): Patients presenting in Emergency Ward of District Hospital, Mustang with AMS (Acute Mountain Sickness), HAPE (High altitude Pulmonary Oedema) or HACE (High altitude Cerebral Oedema) as CASES Healthy volunteers who didn't develop any symptoms of AMS/HAPE/HACE after their trip to high altitude 4.6 Sampling Methods/Techniques (Specify): Random sampling Semi-structured questionnaire will be used for data collection by interview method.

4.7 Sample size (with justification): According to the literature review (6), the prevalence of AMS with rapid ascent was 58% (p1) while with slow ascent was 33% (p2).

The following formula would be used for calculating the adequate sample size in case control study.(13) n=((r+1)p'(1-p^')〖(Z_β+Z_(α/2))〗^2)/(r〖(p1-p2)〗^2 ) Where n is the sample size, Z_β= Standard normal variate for power Z_(α/2)= Standard normal variate for level of significance p1- p2 = Effect size or different in proportion expected based on previous studies. p1 is proportion in cases and p2 is proportion in control.

r= ratio of controls to cases. To be taken as 1 in our study Here, p'=(p1+p2)/2, Z_(α/2)=1.96 (at 95% CI) and Z_β=0.84 (at 80% power) So the calculated value of n= 62.4 The minimum sample size is estimated to be 63 for cases and 63 for controls.

4.8 Criteria for Sample Selection:

Inclusion Criteria:

Cases: Individuals age 18 years or older who have been diagnosed with AMS based on a LLS score of ≥3 or HAPE or HACE.

Controls: Individuals age 18 years or older who did not develop AMS during their trip to high altitude as the cases, and who are matched to cases on age and sex.

Exclusion Criteria :

Those who deny consent for participation. Age<18 years Pregnant Patient

Data Collection Technique / Methods (Specify):

Data will be collected using a structured questionnaire, which will be administered to both cases and controls. The questionnaire will include questions related to demographic characteristics, medical history, exposure history, ascent rate, and symptoms related to high altitude sickness. The questionnaire will be translated into the local language to ensure that participants understand the questions properly.

The questionnaire would comprise two sections: a. Sociodemographic profile of the subject b. Contextual matter which would be studied under different sub headings.

The sociodemographic profile includes Name, Age, Sex, Address and Nationality. Contextual matter comprises basic questions about presenting symptoms at corresponding altitude level of sickness and ascent rate.

Patient presenting with high altitude sickness symptoms will be diagnosed as AMS, HAPE or HACE. If the patient doesn't meet the diagnosis criteria then he/she will not be included in CASES.

AMS will be diagnosed as a Lake Louise AMS score total of three or more points from the four rated symptoms described below, including at least one point from headache in the setting of a recent ascent or gain in altitude. AMS severity assessment will be done according to LLS scoring and will be classified as ; 3-5 = mild, 6-9 = moderate, and 10-12 = severe AMS.(14) Headache 0-None at all

1-A mild headache 2-Moderate headache 3-Severe headache, incapacitating Gastrointestinal symptoms 0-Good appetite

1. Poor appetite or nausea
2. Moderate nausea or vomiting
3. Severe nausea and vomiting, incapacitating Fatigue and/or weakness

0-Not tired or weak

1-Mild fatigue/weakness 2-Moderate fatigue/weakness 3-Severe fatigue/weakness, incapacitating Dizziness/light-headedness 0-No dizziness/light-headedness

1. Mild dizziness/light-headedness
2. Moderate dizziness/light-headedness
3. Severe dizziness/light-headedness, incapacitating HACE will be diagnosed clinically if there is a change in mental status or ataxia in a person with AMS or a change in mental status and ataxia in a person without AMS. For a patient to have HAPE, he or she must have at least two of the following symptoms: dyspnea at rest, cough, weakness or decreased exercise performance, chest tightness or congestion, and at least two of the following signs: crackling sounds or wheezing in at least one lung field, central cyanosis, tachypnea, and tachycardia.(15) *Signs and symptoms occurring in the setting of a recent gain in altitude.

Consent will be taken and English or Nepali Questionnaire will be used according to the compliance of the participants and the pro-forma will be filled.

Sociodemographic profiles will be taken and questions regarding symptoms of presentation, ascent rate, co-morbidities, past history including previous history of altitude sickness, personal History such as smoking, alcohol intake, awareness on High Altitude Sickness and intake of Prophylactic medicine (Acetazolamide).

Controls will be selected from the similar population as the cases, but will not have developed high altitude sickness during their trip. For each case, one control will be selected and matched by age (within two years) and sex.

Controls will be identified from different trekking or mountaineering group as the cases. If a suitable control cannot be found from the same group, controls will be sought from a different group from the same area or time period.

To ensure that the controls have not developed high altitude sickness during the trip, they will be evaluated using the Lake Louise Score or the Environmental Symptoms Questionnaire (ESQ) upon arrival at high altitude and at the end of the trip. Only individuals who did not develop high altitude sickness during the trip will be eligible as controls.

Controls will be interviewed in a similar manner to cases, with questions about demographic information, medical history, ascent rate, medication use, and other factors that may affect the development of high altitude sickness.

The Participants will be expressed gratitude for the effort they have given for the interview.

4.10 Data Collection Tools: (please attached in annex along with participant/case record form): attached pro-forma 4.11 Pre-testing the Data Collection Tools (if relevant): N/A

4.12 Validity and Reliability of the Research (if relevant): Mention, how will you assess validity and reliability?

The following measures were adopted to maintain and increase the reliability and validity of the study:

i. An adequate number of data sets of tools were pre-tested and validity of the tools in its contents and accuracy of information was ensured. In addition, it was believed that the pre-testing had helped increase the understanding of the contents among the research assistants.

ii. Researcher was oriented adequately about administering the tools and its contents in depth before pre-testing.

iii. Review of concerned literatures and opinions from the experts in the concerned field were obtained. Comments from experts were invited and shared with the research tutor throughout the study process.

4.13 Potential Biases (if relevant): Selection bias, Recall Bias 4.14 Limitation of the Study (if relevant): Diagnosis of Acute mountain sickness/HAPE/HACE will be done clinically. No radiological tools will be used.

4.15 Possible Challenges of the Study: Difficulties in Selecting Controls

Plan for Data Management and Statistical Analysis:

Data will be entered in Microsoft Excel and converted it into SPSS for statistical analysis .

Descriptive statistics will be used to summarize the characteristics of cases and controls. Univariate and multivariate logistic regression analyses will be performed to assess the association between risk factors and high altitude sickness. The results will be reported as odds ratios with corresponding 95% confidence intervals. A p-value of less than 0.05 will be considered statistically significant.

Adverse response / side effects reporting: N/A Mention stopping RULES for study: N/A Expected Outcome of the Research: N/A

Plan for Dissemination of Research Results:

Study result will be presented at research meet and also published in national and international indexed journal.

Plan for Utilization of the Research Findings (optional):

Work Plan (should include duration of study, tentative date of starting the project and work schedule / Gantt chart): N/A Ethical Consideration

Regarding the human participants: Human

11.1 Are human participants required in this research? If yes, provide justification.

Yes (provide justification) No

This is descriptive retrospective study done to find out the pattern of presentation of symptoms of Acute mountain sickness

11.2 How many participants are required for the research? Explain. Our study includes patients coming to Emergency in six month study period.

11.3 What is the frequency of the participant's involvement in the research? Explain.

(Follow up the schedule): N/A

11.4 Clearly indicate the participant's responsibilities in the research. What is expected of the research participants during the research? N/A

11.5 Are you studying vulnerable members include - pregnant / newborn / children below 12 years / physically or mentally challenges / HIV / AIDS / IV drug users for this research? If yes, provide justification: No

11.6 Are there any risks involved to the participants? If yes, identify clearly what are the expected risks for the human participants in the research and provide a justification for these risks: N/A

11.7 Are there any benefits involved to the participants? If yes, identify clearly what are the expected benefits for the participants. No

Informed written Consent Form / Ethical Issues (please attach in annex): attached below

ELIGIBILITY:
Inclusion Criteria:

Cases: - Individuals age 18 years or older who have been diagnosed with AMS based on a LLS score of ≥3 or HAPE or HACE.

Controls: - Individuals age 18 years or older who did not develop AMS during their trip to high altitude as the cases, and who are matched to cases on age and sex.

Exclusion Criteria:

* Those who deny consent for participation.
* Age<18 years
* Pregnant Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting in Emergency Ward of District Hospital, Mustang with AMS (Acute Mountain Sickness), HAPE (High altitude Pulmonary Oedema) or HACE (High altitude Cerebral Oedema) as CASES Healthy volunteers who didn't develop any symptoms of AMS/HAPE/HACE after their trip to high altitude
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Ascent Rate | 6 months
Awareness on High Altitude Sickness | 6 months
Personal History such as smoking, alcohol intake, recreational drugs | 6 months
Intake of Prophylactic medicine (Acetazolamide) | 6 months
Past history of Covid-19 , TB | 6 months
Past History including previous history of altitude sickness | 6 months
Co-morbidities | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mustang District Hospital, Jomsom, Gandaki, Nepal

IPD SHARING:
Plan to Share IPD: Undecided